CLINICAL TRIAL: NCT02698865
Title: A Pivotal Study Comparing Two Injections of MONOVISC to Two Injections of Saline in Patients With Osteoarthritis of the Hip
Brief Title: The MONOVISC Hip Osteoarthritis Study
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The results of the interim analysis indicate the futility criterion have been met, therefore enrollment was terminated.
Sponsor: DePuy Mitek (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 15-MVH-01
Record Dates: First submitted 2016-02-25; First posted 2016-03-04 (Estimated); Results first posted 2020-03-04 (Actual); Last update posted 2021-12-01 (Actual); Status verified 2021-11

CONDITIONS: Osteoarthritis of the Hip
MeSH Terms: conditions — Osteoarthritis, Hip

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- MONOVISC (Experimental): MONOVISC High Molecular Weight Hyaluronan
  Interventions: Device: MONOVISC
- Saline (Placebo Comparator): Physiologic saline
  Interventions: Device: Saline

INTERVENTIONS:
Device: MONOVISC — Two (2) intra-articular injections of 4 ml MONOVISC, separated by 1 month, delivered under image guidance (ultrasound or fluoroscopy)
  Arms: MONOVISC
Device: Saline — Two (2) intra-articular injections of 4 ml saline, separated by 1 month, delivered under image guidance (ultrasound or fluoroscopy)
  Arms: Saline

SUMMARY:
This study is being done to determine the effectiveness of MONOVISC for the relief of pain and symptoms of osteoarthritis of the hip. Specifically, the study will determine if MONOVISC is more effective than a placebo treatment when delivered as intra-articular injections (injected directly into the hip joint). In this case, the placebo will be a dilute solution of salt water (saline).

DETAILED DESCRIPTION:
The primary objective of this study is determine whether two intra-articular injections of MONOVISC, separated by 1 month, are superior to two intra-articular injections of physiologic saline, separated by 1 month, in relieving hip osteoarthritis pain, as determined by reduction in walking pain change from baseline.

ELIGIBILITY:
Inclusion Criteria:

* Male or female ≥ 30 years old
* Body Mass Index (BMI) ≤ 35
* Clinical or radiographic diagnosis of hip osteoarthritis in the target hip, with a Kellgren-Lawrence (K/L) grade of 2 or 3.
* Walking pain NRS ≥ 4 and ≤ 8.
* Willing to discontinue all pain medications (except rescue medication) for 7 days prior to the first study injection and for the duration of the study.
* Willing to discontinue rescue medication for 48 hours prior to the first study injection.
* Willing to discontinue rescue medication for 48 hours prior to all follow-up visits
* Ability to tolerate acetaminophen (e.g. Tylenol).
* Must be physically and mentally willing and able to comply with pre and post-treatment scheduled clinical and radiographic evaluations
* Must voluntarily sign the Institutional Review Board approved Informed Consent Form.
* Must agree not to initiate cannabis therapy during the trial study period.

Exclusion Criteria:

* Radiographic evidence of osteonecrosis in the target hip
* NRS walking pain ≥ 3 the contralateral hip
* Clinically diagnosed osteoarthritis in either knee resulting in walking pain greater than NRS 5.
* Dependence on external stabilization for walking (e.g. cane, crutches, walker, etc.)
* Pain associated with lower back disorders that cannot be differentiated from target hip pain
* Major dysplasia or congenital abnormality
* Diagnosis of fibromyalgia
* Primary inflammatory arthropathy, or any other condition affecting the joint, including rheumatoid arthritis or gout in the target hip
* Any musculoskeletal condition that could impede efficacy measurement of the target hip
* Any major surgery, arthroplasty, or arthroscopy of the lower extremities in the past 6 months, or planned surgery during the study
* Infection of the injection site area
* Chronic skin disorders that could interfere with injection site evaluation
* Patients with asthma who require systemic use of corticosteroids
* Septic arthritis in any joint in the past 12 weeks
* For all patients: known hypersensitivity to hyaluronan, lidocaine, or acetaminophen
* For patients undergoing fluoroscopic injection guidance: known hypersensitivity to iodine-based fluoroscopic contrast agents, shellfish, or iodine
* Intra-articular steroid injection of the target hip within the last 3 months or hyaluronan injection of the target hip within the last 26 weeks
* Systemic corticosteroids within the last 12 weeks
* Glucosamine and/or chondroitin sulfate within last 4 weeks
* Currently on anticoagulation therapy, including aspirin therapy of > 81 mg/day (e.g. one daily "baby aspirin").
* Uncontrolled diabetes mellitus.
* Pregnant or breast feeding, or plan to be pregnant during the course of the study
* Any significant illness (metastasis of any type) that decreases the probability of the subject's survival to the 26 week endpoint
* Patients unwilling/unable to complete a pain/function and quality of life questionnaires
* Significant trauma to the index hip within 26 weeks of screening
* Is receiving workman's compensation, or is currently involved in litigation relating to hip osteoarthritis
* Is receiving prescription pain medication for conditions unrelated to hip osteoarthritis
* Chronic use of narcotics
* Unwilling to return for follow-up visits as described in this protocol
* Otherwise determined by the investigator to be medically unsuitable for participation in this study

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2019-03-15 (Actual); Study Completion 2019-06-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brooks J Story, PhD, Study Director — DePuy Synthes Mitek Sports Medicine
Locations (27):
- United States (27):
  - Tucson Orthopedic Institute, Tucson, Arizona
  - CORE Orthopedic Medical Center, Encinitas, California
  - Eisenhower Medical Center/Desert Orthopedic Center, Rancho Mirage, California
  - Southern California Orthopedic Institute, Van Nuys, California
  - University of Colorado - Denver, Denver, Colorado
  - Denver Hip and Knee, Denver, Colorado
  - Center for Arthritis and Rheumatic Diseases, Miami, Florida
  - Integral Rheumatology & Immunology Specialists, Plantation, Florida
  - Emory Sports Complex, Brookhaven, Georgia
  - Iowa Orthopedic Center, Des Moines, Iowa
  - Sports Medicine North, Peabody, Massachusetts
  - MedSport - University of Michigan, Ann Arbor, Michigan
  - Professional Orthopedics, Cherry Hill, New Jersey
  - Hospital for Special Surgery, New York, New York
  - Columbia Medical Center, New York, New York
  - University of North Carolina, Chapel Hill, North Carolina
  - OrthoCarolina Sports Medicine Center, Charlotte, North Carolina
  - Sanford Health, Fargo, North Dakota
  - Cleveland Clinic, Garfield Heights, Ohio
  - Rothman Institute, Media, Pennsylvania
  - Texas Orthopedic Specialists, Bedford, Texas
  - Houston Methodist, Houston, Texas
  - Inov8 Orthopaedics, Houston, Texas
  - San Antonio Orthopaedic Group, San Antonio, Texas
  - University of Virginia, Charlottesville, Virginia
  - National Sports Medicine Institute, Lansdowne Town Center, Virginia
  - OrthoVirginia, Lynchburg, Virginia

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Groups:
- Monovisc: Participants received the intra-articular injections of 4 mL (milliliter) monovisc high molecular weight hyaluronan as active treatment into the hip joint on Day 1 and then second injection on Day 31.
- Saline: Participants received the intra-articular injections of 4 mL (milliliter) physiologic saline as control treatment into the hip joint on Day 1 and then second injection on Day 31.
Period: Overall Study
Arm/Group | Monovisc | Saline
Started | 140 | 80
Treated | 140 | 80
Completed | 105 | 47
Not Completed | 35 | 33
Not completed — Other | 11 | 11
Not completed — Withdrawal by Subject | 20 | 16
Not completed — Physician Decision | 0 | 4
Not completed — Lost to Follow-up | 4 | 2

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set (SAS) consists of all randomized participants who were enrolled in the study and received either Monovisc or Saline and were analyzed as per treatment received.
Groups:
- Total: Total of all reporting groups
Arm/Group | Monovisc | Saline | Total
Number analyzed (Participants) | 140 | 80 | 220
Age, Continuous [Mean (Standard Deviation); unit: Years] | 58.5 (9.55) | 59.4 (10.80) | 58.8 (10.01)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 84 | 46 | 130
  Male | 56 | 34 | 90
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 20 | 10 | 30
  Not Hispanic or Latino | 120 | 70 | 190
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 6 | 3 | 9
  White | 133 | 75 | 208
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Walking Pain as Measured by Western Ontario and McMaster Universities Arthritis Index (WOMAC) A1 Score at Day 180
Description: The Western Ontario and McMaster Universities Arthritis Index (WOMAC) is widely used in the evaluation of Hip and Knee Osteoarthritis. Walking Pain Score is measured by question A1 on the WOMAC 3.1 Index. The WOMAC questionnaire used in this study was administered in the Numerical rating scale (NRS) format. Question A1 on the WOMAC 3.1 Index measures the amount of pain that a participant has when walking on a flat surface. It is one question that is collected on a scale from 0 to 10 where a score of 0 indicates no pain and a score of 10 indicates extreme pain.
Time Frame: Baseline and Day 180
Population: Safety Analysis Set (SAS) consists of all randomized participants who were enrolled in the study and received either Monovisc or Saline and were analyzed as per treatment received. Here 'N' (number of participants analyzed) signifies participants who were evaluable for this outcome measure (OM).
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Monovisc | Saline
Number analyzed (Participants) | 105 | 47
Units on a scale | -1.75 (2.88) | -1.53 (3.21)

2. Secondary Outcome: Change From Baseline in Walking Pain as Measured by Western Ontario and McMaster Universities Arthritis Index (WOMAC) A1 Score at Day 14, 28, 60 and 120
Description: as for outcome 1
Time Frame: Baseline, Day 14, 28, 60 and 120
Population: SAS consists of all randomized participants who were enrolled in the study and received either Monovisc or Saline and were analyzed as per treatment received. Here 'n'(number analyzed) signifies participants who were evaluable at specified timepoints.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Monovisc | Saline
Number analyzed (Participants) | 140 | 80
Units on a scale
  Change at Day 14: number analyzed (Participants) | 137 | 76
  Change at Day 14 | -1.44 (2.32) | -1.16 (2.14)
  Change at Day 28: number analyzed (Participants) | 130 | 71
  Change at Day 28 | -1.42 (2.46) | -1.13 (2.19)
  Change at Day 60: number analyzed (Participants) | 122 | 68
  Change at Day 60 | -1.89 (2.76) | -1.75 (2.31)
  Change at Day 120: number analyzed (Participants) | 113 | 53
  Change at Day 120 | -1.97 (2.79) | -1.58 (2.8)

ADVERSE EVENTS:
Time Frame: Up to 36 months
Description: Safety Analysis Set (SAS) consisted of all randomized participants who were enrolled in the study and received either Monovisc or Saline and were analyzed as per treatment received.
Arm/Group | Monovisc | Saline
All-Cause Mortality (participants affected / at risk) | 0/140 | 0/80
Serious Adverse Events (participants affected / at risk) | 2/140 | 0/80
Other Adverse Events (participants affected / at risk) | 25/140 | 12/80
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Monovisc (N=140) | Saline (N=80)
Mitral Valve Prolapse (Cardiac disorders) | 1 | 0
Hip Arthroplasty (Surgical and medical procedures) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Monovisc (N=140) | Saline (N=80)
Arthralgia (Musculoskeletal and connective tissue disorders) | 25 | 12

LIMITATIONS AND CAVEATS:
No Study limitation was reported for this study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation. If requested in writing, such publication will be withheld for up to an additional 60 days.

DOCUMENTS (2):
  • Study Protocol (2017-10-30): https://cdn.clinicaltrials.gov/large-docs/65/NCT02698865/Prot_000.pdf
  • Statistical Analysis Plan (2016-03-01): https://cdn.clinicaltrials.gov/large-docs/65/NCT02698865/SAP_001.pdf